CLINICAL TRIAL: NCT04763629
Title: Comparative Effects on Short-term Blood Pressure Variability and Left Atrial Function of Interval Combined Training Versus Continuous Combined Training in Hypertensive Patents With Ischemic Heart Disease.
Brief Title: Effects of Different Exercise Training Programs on Short-term Blood Pressure Variability and Atrial Function in Hypertension
Acronym: TACITO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele Roma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RP 21/28
Record Dates: First submitted 2021-02-18; First posted 2021-02-21 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Hypertension; Coronary Artery Disease
Keywords: atrial function; hypertension; coronary artery disease
MeSH Terms: conditions — Hypertension; Coronary Artery Disease | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interval Combined Training (ICT) (Experimental): Patients randomized to this group will perform aerobic exercise on the stationary cycle ergometer using an interval protocol consisting of alternating bouts of 5 minutes at 80-90% of VO₂ peak and 10 minutes at 50-60% of VO₂ peak. This sequence will be repeated three times, resulting in a total aerobic exercise duration of 45 minutes. Then they will perform dynamic resistance exercise lasting 35 minutes at 60% of 1-repetition maximum (1-RM)
  Interventions: Other: Physical exercise
- Continuous Combined Training (CCT) (Experimental): Patients randomized to this group will perform 45 minutes of cycling at a constant heart rate corresponding to 60-70% of VO₂ peak as determined during cardiopulmonary test. Then they will perform dynamic resistance exercise at 60% of 1-RM involving arms and legs for 35 minutes.
  Interventions: Other: Physical exercise

INTERVENTIONS:
Other: Physical exercise — Patients of both arms will undergo two different modalities of exercise during the 12 weeks study period.

SUMMARY:
The study aim is to compare the effects produced by two different exercise training modalities on short-term blood pressure variability and atrial function evaluated by speckle-tracking echocardiography in hypertensive patients with ischemic heart disease. 50 males patients will be randomized to interval combined training (ICT) o0r aerobic continuous combined training (CCT) botrg including aerobic and resistance exercises. The training period will last 12 weeks. The protocol will provide two different assessment of atrial function: -acute: after a single session of exercise; - 12 weeks: at the end of exercise training protocols. 24/h blood pressure variability will be performed before starting the training programs and at 12 weeks.

DETAILED DESCRIPTION:
This is a prospective randomized two- arms, single-blinded, parallel trial evaluating the effects of two different exercise training modalities on atrial function, assessed by speckle-tracking echocardiography, and shortt-term blood pressure variability in hypertensive patients with coronary artery disease. First endpoint will be: between-groups comparison of changes in short-term BP variability. Secondary endpoints will be: exercise-induced changes in peak atrial longitudinal strain (PALS); diastolic function, left ventricular strain, 24/h blood pressure values, exercise tolerance. We will include 50 patient with hypertension and underlying coronary artery disease, evaluated for entering a cardiac rehabilitation program. Patients that will be judged suitable for the study will be randomized, with a 1:1 ratio, to interval combined training (ICT) or aerobic continuous combined training (CCT) both including aerobic and resistance exercises. Each patient will undergo three visits. At visit 1 in which patients will perform a first echocardiography with evaluation of the acoustic window and a cardiopulmonary test (for excluding myocardial ischemia and for establishing the training intensity); visit 2- acute evaluation- :patients will undergo an echocardiographic assessment before and within 30 minutes after a single exercise session (alternatively interval or combined training according to the randomization code). Visit 3: at 12 weeks all patient will perform a final echocardiography evaluation, a 24/h blood pressure monitoring and a second cardiopulmonary test. Patients of both groups will exercise three times/week for 12 weeks. Each exercise session will last 80 minutes

ELIGIBILITY:
Inclusion Criteria:

* Hypertension;
* Coronary artery disease;
* Age over 45 years;
* Male gender

Exclusion Criteria:

* Secondary hypertension;
* Significant heart valve diseases;
* Hypertrophic cardiomyopathy;
* Signs and/or symptoms of myocardial ischemia during an ergometric test;
* Uncontrolled arrhythmia;
* Neurological and or orthopedic conditions contraindicating or limiting exercises;
* Significant chronic obstructive pulmonary disease (FEV1 <50%),
* Symptomatic peripheral arterial disease

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 40 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
changes on peak atrial longitudinal strain | 12 weeks
  between-groups comparison of exercise-induced changes on peak atrial longitudinal strain

SECONDARY OUTCOMES:
changes on left ventricle global longitudinal strain | 12 weeks
  between-groups comparison of exercise-induced changes on left ventricle global longitudinal strain

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Caminiti, Study Chair — IRCCS San Raffaele Rome
Locations (1):
- IRCCS San Raffaele Pisana, Rome, Italy